CLINICAL TRIAL: NCT01745991
Title: Randomised Control Trial to Investigate the Effectiveness of CoSeal® Surgical Sealant in Reducing Intra-abdominal Adhesions Following the Kasai Hepatoportoenterostomy for Biliary Atresia.
Brief Title: Trail to Investigate the Effectiveness of CoSeal in Reducing Adhesions Following the Kasai Hepatoportoenterostomy for Biliary Atresia
Acronym: CoSRCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Naved Alizai (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, Naved Alizai, Consultant Paediatric Surgeon, The Leeds Teaching Hospitals NHS Trust
Organization: The Leeds Teaching Hospitals NHS Trust (Other)
Other Study IDs: NKA/LTHT/UK/CoSealRCT
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biliary Atresia undergoing Kasai op: Randomisation for the use of CoSeal at the time of Kasai and assessment at the time of Transplantation.
  Interventions: Device: CoSeal spray

INTERVENTIONS:
Device: CoSeal spray

SUMMARY:
The investigators plan to invite all children in the UK with biliary atresia, treated at the three national centres (Birmingham, Kings College and Leeds), over a three year period to take part in a randomised control study. The investigators aim to determine the effectiveness of CoSeal® Surgical Sealant (an anti-adhesive agent) in reducing intra-abdominal adhesions (scar tissue) and the morbidity caused by these adhesions in children treated with a Kasai hepatoportoenterostomy. Adhesions are common, if not invariable, after any abdominal surgery. They cause intra-abdominal organs to become stuck to each other and the abdominal wall. This means they are no longer completely free to slide over each other. In particular patients have a lifetime risk that the bowel can become kinked or twisted leading to complications such as bowel obstruction. Adhesions also make repeat abdominal operations more difficult. The adhesions have to be divided in order to separate the organs from each other and the abdominal wall. This can lead to blood loss and increases the risk of damage to these organs. Anti-adhesive agents have been created to reduce the severity of these adhesions, but there is little in the medical literature to evaluate their effectiveness, particularly in children. Biliary atresia is an obliterative obstruction of the bile ducts that occurs in infants. Initially they are treated by an abdominal operation called a Kasai portoenterostomy to restore bile flow from the liver to the intestines. However approximately 40% of these children will go on to require a liver transplant operation in the first two years of life. If CoSeal® Surgical Sealant is effective this could reduce the patients lifetime risk of complications from abdominal adhesions and also facilitate repeat abdominal operations for these children, in particular for those who go on to require a liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Biliary Atresia undergoing Kasai Hepatoportoenterostomy.

Exclusion Criteria:

* Patients with BA and malrotation

Ages: 7 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 126 patients over a three year period
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Severity of Intra-abdominal adhesions | 5 years
  Adhesions assessed at the time of Liver transplantation

SECONDARY OUTCOMES:
Liver transplantation- blood loss | 5 years
Liver Transplantation- Time taken | 5 years

OTHER OUTCOMES:
Bowel damage | 5 years
Intra-abdominal sepsis | 5 years
Re-operation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Naved Alizai, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (3):
- United Kingdom (3):
  - Leeds General Infirmary, Leeds, West Yorkshire
  - Khalid Sharif, Birmingham Children's Hospital
  - Mark Davenport, Kings College Hospital, London